CLINICAL TRIAL: NCT02837315
Title: Improving Brief Marijuana Interventions With a Behavioral Economic Supplement
Acronym: BLUE-J
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, James G Murphy, Professor, University of Memphis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3R01AA020829-02S1 (NIH); 4R01AA020829-05 (NIH)
Record Dates: First submitted 2016-07-11; First posted 2016-07-19 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Marijuana Use
MeSH Terms: conditions — Marijuana Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BMI + SFAS (Experimental): Participants first receive a 50-minute standard brief motivational intervention designed to reduce marijuana use. A week later, they will receive the SFAS (Substance-free Activity Session., a 50-minute counseling session designed to increase the salience of the student's academic and career goals, draw attention to the potentially negative relationship between substance use and goal accomplishment, and increase engagement in substance-free alternative activities. The SFAS was described to participants as the "College Adjustment Session" and the session was conducted using an MI plus personalized feedback approach.
  Interventions: Behavioral: Brief Motivational Intervention (BMI); Behavioral: Substance-Free Activity Session (SFAS)
- BMI + Relaxation Session (Active Comparator): Participants first receive a 50-minute standard brief motivational intervention designed to reduce marijuana use. A week later, they will receive a relaxation training session. In the relaxation training session, the clinician leads the student through a diaphragmatic breathing exercise, followed by a progressive muscle relaxation protocol (~30 minutes). At the end of the session, students were asked about their reaction to the relaxation techniques and were provided with relaxation training handouts.
  Interventions: Behavioral: Brief Motivational Intervention (BMI); Behavioral: Relaxation Session
- Assessment (No Intervention): Participants fill out a battery of measures and receive no intervention.

INTERVENTIONS:
Behavioral: Brief Motivational Intervention (BMI) — This session includes a discussion related to harm reduction and the student's autonomy to make decisions about the information provided in the session; a marijuana use decisional balance exercise; personalized marijuana-related feedback, and goal-setting. Elements included in the feedback are: (a) comparison of the student's perception of how much college students use marijuana and actual student norms, (b) a comparison of the student's marijuana use vs. norms, (c) drug-related problems experienced, (e) money spent on marijuana, and (f) alcohol norms and consequences if participants indicated they also drink alcohol. Participants discuss the personalized feedback with the clinician and review protective behavioral strategies if she or she indicates interest.
  Arms: BMI + Relaxation Session; BMI + SFAS
Behavioral: Substance-Free Activity Session (SFAS) — The clinician initiates a discussion of the student's college and career goals. Students discuss the values that motivate them as well as how marijuana use may interfere with their ability to accomplish these goals. Students then receive information on graduation rates and income benefits for those who attend and excel in college. They receive personalized feedback on (a) the requirements for their major and intended career, (b) a list of extracurricular activities tailored to their goals, (c) a graph showing time they allocate to their activities, (d) information on stress and depressive symptoms (if applicable) and possible adaptive coping responses and (e) a list of substance-free recreational activities in which they would like to start or continuing engaging.
  Arms: BMI + SFAS
Behavioral: Relaxation Session — The session includes a clinician-led diaphragmatic breathing exercise, followed by a progressive muscle relaxation protocol (~30 minutes). At the end of the session, students are asked about their reaction to the relaxation techniques and are provided with relaxation training handouts.
  Arms: BMI + Relaxation Session

SUMMARY:
The purpose of this study is to evaluate the efficacy of a Substance-Free Activity Session (SFAS) as a supplement to a brief motivation intervention (BMI) in reducing marijuana use and drug-related consequences in college student

DETAILED DESCRIPTION:
Approximately 20% of college students are regular marijuana users, and are at risk for cognitive and academic problems, addiction, and risk behaviors such as driving while impaired. Young adult marijuana users are thus a high-risk population and may require an intervention that motivates marijuana reductions by increasing engagement in constructive alternatives to marijuana use. Brief Motivational Interventions (BMIS) have demonstrated efficacy for alcohol use in college students, but lack consistent evidence of efficacy for marijuana use. This research team has developed a supplement to alcohol BMIs, the Substance-Free Activity Session (SFAS), which directly targets the behavioral economic mechanisms of both substance-free reinforcement and delayed reward discounting by encouraging the development of and commitment to academic and career goals, and by highlighting the impact of day-to-day patterns of alcohol use and academic engagement on these goals. A controlled pilot trial found that the SFAS improved BMI outcomes in a sample of heavy drinking college students, and the ongoing parent trial to this revision is replicating and extending those results. This study will evaluate the SFAS using a randomized 3-group (BMI + SFAS vs. BMI + Relaxation Attention Control, vs. Assessment Only) pilot trial with 120 undergraduates (50% female, 40% minority) who report using marijuana on > 5 days in the past-month. It is hypothesized that at the 1-month and the next-semester follow-ups (follow-ups are wedded to the academic calendar to allow for representative measurement of marijuana use and activity patterns) BMI+SFAS participants will report significantly lower levels of marijuana use and problems, and that these reductions will exceed those of BMI + Relaxation and Assessment-Only participants. Exploratory analyses will test the hypotheses that (a) the BMI + SFAS will be more effective for participants who report higher baseline marijuana reinforcing efficacy and delayed reward discounting; and (b) the advantage of BMI + SFAS on marijuana use will be mediated by increased participation in substance-free activities. Support for our hypotheses would extend behavioral economic theory and would provide initial validation for an approach that could be used to reduce marijuana misuse among the increasing population of college students who misuse marijuana. Furthermore, given the focus of the SFAS is to increase academic/campus engagement, this work has the potential for widespread dissemination.

ELIGIBILITY:
Inclusion Criteria:

* freshman or sophomore at the university of Memphis
* 5 or more past-month days of marijuana use

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Marijuana use | Baseline, 1-month, 6-months
  Electronic timeline follow-back to measure marijuana use days

CONTACTS AND LOCATIONS:
Overall Officials: James G Murphy, Ph.D., Principal Investigator — University of Memphis
Locations (1):
- University of Memphis, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers will maintain a de-identified database and after publishing the primary outcomes, they will make individual level data available to researchers who are conducting integrated analyses.

REFERENCES:
- [Derived] Murphy JG, Dennhardt AA, Utzelmann B, Borsari B, Ladd BO, Martens MP, White HR, Yurasek AM, Campbell KW, Witkiewitz K. A pilot trial of a brief intervention for cannabis use supplemented with a substance-free activity session or relaxation training. Psychol Addict Behav. 2024 May;38(3):255-268. doi: 10.1037/adb0000988. Epub 2024 Jan 25. PMID 38271079